CLINICAL TRIAL: NCT00376376
Title: Urinary Bactericidal Activity of 4 Doses of Levofloxacin (250, 500, &750, and 1000 mg) Against Fluoroquinolone-Resistant E. Coli
Brief Title: Urinary Bactericidal Activity of 4 Doses of Levofloxacin Against Fluoroquinolone-Resistant E. Coli
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MSU 06-496F
Record Dates: First submitted 2006-09-13; First posted 2006-09-14 (Estimated); Last update posted 2008-11-27 (Estimated); Status verified 2008-11

CONDITIONS: Healthy Volunteers
Keywords: levofloxacin; pharmacodynamic; bactericidal

INTERVENTIONS:
Drug: levofloxacin at 250, 500, 750, and 1000 mg doses

SUMMARY:
Single-dose studies of a fluoroquinolone are indicative of their antimicrobial activity since little accumulation occurs with multiple doses. Single-dose studies have been utilized to determine drug concentrations and time kill activity in serum, urine, and respiratory tissues.

The purpose of this study is to evaluate the Urine Bactericidal Activity (UBA) of levofloxacin (250, 500, 750, and 1000 mg) against FQ-resistant, ESBL positive E. coli isolates. In addition, a susceptibility breakpoint concentration in the urine can also be established for each dose of levofloxacin. Furthermore, urine concentrations and serum pharmacokinetic parameters of levofloxacin can be determined.

DETAILED DESCRIPTION:
Subjects: -10 healthy (from medical history) adult male or female volunteers

* Normal body weight (within 20 %)
* Age range: 18-60
* Not taking any other restricted medications (ie. antibiotics)

Drug : all drugs are a single dose given after a 12 hour fast

* 1000 mg.levofloxacin
* 750 mg. levofloxacin
* 500 mg levofloxacin
* 250 mg levofloxacin

Levofloxacin Pharmacokinetic Study:

A serum sample will be obtained prior to and at 1.5 (peak), 4.0, 8.0, 12 (50% of interval) and 24 (100% of interval) hours after each single dose of levofloxacin (6 time points).

Levels will be determined by an HPLC assay.

Urine Pharmacodynamic Study:

A urine sample will be obtained prior to and at 1.5 (peak), 4, 8, 12 (50% of interval), and 24 (100% of interval) hours after a single dose of each dose of levofloxacin.

A urine pH will be run on each sample.

All urine levels will be determined by a validated HPLC assay.

Study Isolates: E. coli (TRUST isolates):

Levofloxacin MICs:

* 0.125 (sensitive)
* 4.0 (intermediate)
* 8.0 (resistant)
* 16.0 (resistant)
* 32.0 (resistant)
* 64.0 (resistant)

This MIC range of E. coli isolates should be able to define a levofloxacin susceptibility breakpoint for urinary pathogens at each dose studied.

Urine Cidal Activity: Urine samples will be tested against each of the study isolates. A maximum urine cidal titer will be determined for each urine. The median titer at each time period (10 subjects) will determine the urine cidal activity.

The duration of cidal activity for each isolate will be determined and plotted. A 12-h duration will be considered the minimum time necessary for prolonged Urine Bactericidal Activity (MIC breakpoints).

Safety: All patients will be monitored for side effects during the study.

ELIGIBILITY:
Inclusion Criteria:

* healthy (from medical history) adult male or female volunteers
* Normal body weight (within 20 %)
* Age range: 18-60
* Not taking any other restricted medications (ie. antibiotics)

Exclusion Criteria:

* Non-healthy volunteers
* pregnant women
* volunteers on other antibiotics
* body weight over 20% of normal
* Age <18 or >60

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10
Dates: Start 2006-09; Study Completion 2006-11

PRIMARY OUTCOMES:
evaluate the Urine Bactericidal Activity (UBA) of different doses and urine levels of levofloxacin against drug-resistant bacteria.

CONTACTS AND LOCATIONS:
Overall Officials: Gary E. Stein, Pharm.D., Principal Investigator — Michigan State University; Daniel Havlichek, M.D., Principal Investigator — Michigan State University
Locations (1):
- Michigan State University- Dept. of Medicine, East Lansing, Michigan, United States